CLINICAL TRIAL: NCT00801216
Title: High-dose Sequential Chemotherapy and Rituximab (R-HDS) in Patients With Systemic B-cell Lymphoma With Central Nervous System Involvement at Diagnosis or Relapse
Brief Title: High-dose Sequential Chemoimmunotherapy for B-cell Lymphomas With Central Nervous System Involvement
Acronym: SCNSL1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrés José Maria Ferreri (Other)
Collaborators: Mundipharma Pte Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Andrés José Maria Ferreri, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCNSL1; 2006-006999-38 (EudraCT Number)
Record Dates: First submitted 2008-11-28; First posted 2008-12-03 (Estimated); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: B-cell Lymphomas
Keywords: B-cell lymphomas; lymphomatous meningitis; liposomal cytarabine; autologous transplant; CNS involvement; Secondary CNS lymphomas
MeSH Terms: conditions — Lymphoma, B-Cell; Meningeal Carcinomatosis | interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High-dose sequential chemoimmunotherapy (Experimental): Two courses of methotrexate 3.5 g/mq day 1 and cytarabine 2 g/mq twice a day, for two days, Rituximab 375 mg/mq days 3 & 11 and Intrathecal liposomal cytarabine 50 mg day 6(Phase I) followed in case of response by cyclophosphamide 7 g/mq plus Rituximab 375 mg/mq and Intrathecal liposomal cytarabine 50 mg Leukapheresis A and cryopreservation (Phase II), Cytarabine 2 g/mq twice a day for 4 days, Rituximab 375 mg/m2 and Reinfusion of stem cells (Phase III), etoposide 2 g/mq, Intrathecal liposomal cytarabine 50 mg (Phase IV) and high-dose Thiotepa-BCNU supported by autologous stem cell transplant (Phase V), and whole-brain radiotherapy in patients who do not achieve a complete remission after chemotherapy (Phase VI)
  Interventions: Drug: High-dose sequential chemotherapy and autologous transplant

INTERVENTIONS:
Drug: High-dose sequential chemotherapy and autologous transplant — Two courses of methotrexate 3.5 g/mq day 1 and cytarabine 2 g/mq twice a day, for two days, Rituximab 375 mg/mq days 3 & 11 and Intrathecal liposomal cytarabine 50 mg day 6(Phase I) followed in case of response by cyclophosphamide 7 g/mq plus Rituximab 375 mg/mq and Intrathecal liposomal cytarabine 50 mg Leukapheresis A and cryopreservation (Phase II), Cytarabine 2 g/mq twice a day for 4 days, Rituximab 375 mg/m2 and Reinfusion of stem cells (Phase III), etoposide 2 g/mq, Intrathecal liposomal cytarabine 50 mg (Phase IV) and high-dose Thiotepa-BCNU supported by autologous stem cell transplant (Phase V), and whole-brain radiotherapy in patients who do not achieve a complete remission after chemotherapy (Phase VI)
  Other Names: Depocyte

SUMMARY:
This prospective trial will assess the activity and feasibility of a new high-dose methotrexate-based high-dose sequential chemotherapy combination in patients with B-cell lymphomas and CNS involvement at diagnosis or relapse. Selected drugs, with a well-documented anti-lymphoma activity, will be administered at high doses to increase blood-brain barrier penetration and CNS bioavailability as well as to reduce potential cross-resistance.

DETAILED DESCRIPTION:
Patients with aggressive B-cell lymphoma and involvement of the central nervous system at diagnosis or relapse will be treated with a combination of high-dose methotrexate and high-dose cytarabine, rituximab, and intrathecal depocyte followed by rituximab-high-dose sequential chemotherapy supported by autologous tsem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of diffuse large-cell, follicular or mantle cell lymphoma
2. CNS involvement (brain, meninges, cranial nerves, eyes, and/or spinal cord) at diagnosis or relapse after conventional chemotherapy
3. Diagnosis of CNS involvement either by brain biopsy or CSF cytology examination. Neuroimaging alone is acceptable only when stereotactic biopsy is formally contraindicated.
4. Age 18-70 years
5. ECOG performance status 0-3
6. Adequate bone marrow (PLT > 100000 mm3, Hb > 9 g/dl, ANC > 2.000 mm3), renal (creatinine clearance > 60 mL/min), cardiac (VEF > 50%), and hepatic function (total serum bilirubin < 3 mg/dL, AST/ALT and gammaGT < 2.5 per upper normal limit value), within 1 week prior to study start (unless the abnormality is due to lymphoma involvement)
7. Absence of symptomatic coronary artery disease, cardiac arrhythmias not well controlled with medication or myocardial infarction within the last 6 months (New York Heart Association Class III or IV heart disease)
8. Absence of HIV infection
9. No previous or concurrent malignancies with the exception of surgically cured carcinoma in-situ of the cervix and carcinoma of the skin and of other cancers without evidence of disease at least from 5 years
10. Absence of any familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
11. Female patients must be non-pregnant and non-lactating. Sexually active patients of childbearing potential must implement adequate contraceptive measures during study participation
12. No treatment with other experimental drugs within the 6 weeks previous to enrolment
13. Give written informed consent prior to any study specific procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice

Exclusion Criteria:

* NA

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrés J. Ferreri, MD, Study Chair — San Raffaele Scientific Institute
Locations (1):
- San Raffaele Scientific Institute, Milan, Italy

REFERENCES:
- [Derived] Ferreri AJ, Donadoni G, Cabras MG, Patti C, Mian M, Zambello R, Tarella C, Di Nicola M, D'Arco AM, Doa G, Bruno-Ventre M, Assanelli A, Foppoli M, Citterio G, Fanni A, Mule A, Caligaris-Cappio F, Ciceri F. High Doses of Antimetabolites Followed by High-Dose Sequential Chemoimmunotherapy and Autologous Stem-Cell Transplantation in Patients With Systemic B-Cell Lymphoma and Secondary CNS Involvement: Final Results of a Multicenter Phase II Trial. J Clin Oncol. 2015 Nov 20;33(33):3903-10. doi: 10.1200/JCO.2015.61.1236. Epub 2015 Aug 17. PMID 26282634
- See also: Intergruppo Italiano Linfomi web site — https://filinf.it/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 patients were registered, but only 38 patients met the inclusion critaria and was treatted
Groups:
- High-dose Sequential Chemoimmunotherapy: Two courses of methotrexate 3.5 g/mq day 1 and cytarabine 2 g/mq twice a day, for two days, Rituximab 375 mg/mq days 3 & 11 and Intrathecal liposomal cytarabine 50 mg day 6(Ph I) followed in case of response by cyclophosphamide 7 g/mq plus Rituximab 375 mg/mq and Intrathecal liposomal cytarabine 50 mg Leukapheresis A and cryopreservation (Ph II), Cytarabine 2 g/mq twice a day for 4 days, Rituximab 375 mg/m2 and Reinfusion of stem cells (Ph III), etoposide 2 g/mq, Intrathecal liposomal cytarabine 50 mg (Phase IV) and high-dose Thiotepa-BCNU supported by autologous stem cell transplant (Phase V), and whole-brain radiotherapy in patients who do not achieve a complete remission after chemotherapy (Phase VI). High-dose sequential chemotherapy and autologous transplant: Two courses of methotrexate 3.5 g/mq day 1 and cytarabine 2 g/mq twice a day, for two days, Rituximab 375 mg/mq days 3 & 11 and Intrathecal liposomal cytarabine 50 mg day 6(Ph I) followed in case of response by cyclophosphamide 7 g/mq plus Rituximab 375 mg/mq and Intrathecal liposomal cytarabine 50 mg Leukapheresis A and cryopreservation (Ph II), Cytarabine 2 g/mq twice a day for 4 days, Rituximab 375 mg/m2 and Reinfusion of stem cells (Ph III), etoposide 2 g/mq, Intrathecal liposomal cytarabine 50 mg (Ph IV) and high-dose Thiotepa-BCNU supported by autologous stem cell transplant (Phase V), and whole-brain radiotherapy in patients who do not achieve a complete remission after chemotherapy (Phase VI)
Period: Overall Study
Arm/Group | High-dose Sequential Chemoimmunotherapy
Started | 40
Completed | 38
Not Completed | 2
Not completed — Screening Failure | 2

BASELINE CHARACTERISTICS:
Groups:
- High-dose Sequential Chemoimmunotherapy: Two courses of methotrexate 3.5 g/mq day 1 and cytarabine 2 g/mq twice a day, for two days, Rituximab 375 mg/mq days 3 & 11 and Intrathecal liposomal cytarabine 50 mg day 6(Ph I) followed in case of response by cyclophosphamide 7 g/mq plus Rituximab 375 mg/mq and Intrathecal liposomal cytarabine 50 mg Leukapheresis A and cryopreservation (Ph II), Cytarabine 2 g/mq twice a day for 4 days, Rituximab 375 mg/m2 and Reinfusion of stem cells (Phase III), etoposide 2 g/mq, Intrathecal liposomal cytarabine 50 mg (Ph IV) and high-dose Thiotepa-BCNU supported by autologous stem cell transplant (Phase V), and whole-brain radiotherapy in patients who do not achieve a complete remission after chemotherapy (Ph VI)
  High-dose sequential chemotherapy and autologous transplant: Two courses of methotrexate 3.5 g/mq day 1 and cytarabine 2 g/mq twice a day, for two days, Rituximab 375 mg/mq days 3 & 11 and Intrathecal liposomal cytarabine 50 mg day 6(Phase I) followed in case of response by cyclophosphamide 7 g/mq plus Rituximab 375 mg/mq and Intrathecal liposomal cytarabine 50 mg Leukapheresis A and cryopreservation (Phase II), Cytarabine 2 g/mq twice a day for 4 days, Rituximab 375 mg/m2 and Reinfusion of stem cells (Phase III), etoposide 2 g/mq, Intrathecal liposomal cytarabine 50 mg (Phase IV) and high-dose Thiotepa-BCNU supported by autologous stem cell transplant (Phase V), and whole-brain radiotherapy in patients who do not achieve a complete remission after chemotherapy (Phase VI)
Arm/Group | High-dose Sequential Chemoimmunotherapy
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] — Some subject as been included with age over 65 years with Promoter approvation thanks to positive clinical evaluation
  years | 59 [36 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 23
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 38

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: No new pathological events in a 2 ys follow-up period
Time Frame: 2-year
Population: No Event registered at a 2ys follow-up of the population included
Measure: Count of Participants; unit: Participants
Groups:
- High-dose Sequential Chemoimmunotherapy: Two courses of methotrexate 3.5 g/mq day 1 and cytarabine 2 g/mq twice a day, for two days, Rituximab 375 mg/mq days 3 & 11 and Intrathecal liposomal cytarabine 50 mg day 6(PH I) followed in case of response by cyclophosphamide 7 g/mq plus Rituximab 375 mg/mq and Intrathecal liposomal cytarabine 50 mg Leukapheresis A and cryopreservation (Phase II), Cytarabine 2 g/mq twice a day for 4 days, Rituximab 375 mg/m2 and Reinfusion of stem cells (Ph III), etoposide 2 g/mq, Intrathecal liposomal cytarabine 50 mg (Ph IV) and high-dose Thiotepa-BCNU supported by autologous stem cell transplant (Phase V), and whole-brain radiotherapy in patients who do not achieve a complete remission after chemotherapy (Phase VI)
  High-dose sequential chemotherapy and autologous transplant: Two courses of methotrexate 3.5 g/mq day 1 and cytarabine 2 g/mq twice a day, for two days, Rituximab 375 mg/mq days 3 & 11 and Intrathecal liposomal cytarabine 50 mg day 6(Phase I) followed in case of response by cyclophosphamide 7 g/mq plus Rituximab 375 mg/mq and Intrathecal liposomal cytarabine 50 mg Leukapheresis A and cryopreservation (Phase II), Cytarabine 2 g/mq twice a day for 4 days, Rituximab 375 mg/m2 and Reinfusion of stem cells (Phase III), etoposide 2 g/mq, Intrathecal liposomal cytarabine 50 mg (Phase IV) and high-dose Thiotepa-BCNU supported by autologous stem cell transplant (Phase V), and whole-brain radiotherapy in patients who do not achieve a complete remission after chemotherapy (Phase VI)
Arm/Group | High-dose Sequential Chemoimmunotherapy
Number analyzed (Participants) | 38
Participants | 16

2. Secondary Outcome: Time to Progression (TTP)
Description: Time elapsed from Lymphoma diagnosis and CNS involvement
Time Frame: 2-year
Measure: Median (Full Range); unit: Months
Groups:
- High-dose Sequential Chemoimmunotherapy: Two courses of methotrexate 3.5 g/mq day 1 and cytarabine 2 g/mq twice day, for two days, Rituximab 375 mg/mq days 3 & 11, Intrathecal liposomal cytarabine 50 mg day 6(Phase I) followed in case of response by cyclophosphamide 7 g/mq plus Rituximab 375 mg/mq and Intrathecal liposomal cytarabine 50 mg Leukapheresis A and cryopreservation (Phase II), Cytarabine 2 g/mq twice a day for 4 days, Rituximab 375 mg/m2 and Reinfusion of stem cells (Phase III), etoposide 2 g/mq, Intrathecal liposomal cytarabine 50 mg (Phase IV) and high-dose Thiotepa-BCNU supported by autologous stem cell transplant (Phase V), and whole-brain radiotherapy in patients who do not achieve a complete remission after chemotherapy (Phase VI) High-dose sequential chemotherapy and autologous transplant: Two courses of methotrexate 3.5 g/mq day 1 and cytarabine 2 g/mq twice a day, for two days, Rituximab 375 mg/mq days 3 & 11 and Intrathecal liposomal cytarabine 50 mg day 6(Phase I) followed in case of response by cyclophosphamide 7 g/mq plus Rituximab 375 mg/mq and Intrathecal liposomal cytarabine 50 mg Leukapheresis A and cryopreservation (Phase II), Cytarabine 2 g/mq twice a day for 4 days, Rituximab 375 mg/m2 and Reinfusion of stem cells (Phase III), etoposide 2 g/mq, Intrathecal liposomal cytarabine 50 mg (Phase IV) and high-dose Thiotepa-BCNU supported by autologous stem cell transplant (Phase V), and whole-brain radiotherapy in patients who do not achieve a complete remission after chemotherapy (Phase VI)
Arm/Group | High-dose Sequential Chemoimmunotherapy
Number analyzed (Participants) | 38
Months | 1 [0 to 69]

3. Secondary Outcome: Overall Survival
Description: Patients alive after 5 years long follow-up
Time Frame: 5 Years
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose Sequential Chemoimmunotherapy
Number analyzed (Participants) | 38
Participants | 16

4. Secondary Outcome: Tolerability OF THE TREATMENT
Description: For the 38 patients enrolled the number of chemotherapy administered / expected during treatment period
Time Frame: 2-year
Population: Number of Chemotherapy cycles planned
Measure: Number; unit: Number of Chemotherapy cycles
Units Other Than Participants: Chemotherapy Expected
Arm/Group | High-dose Sequential Chemoimmunotherapy
Number analyzed (Participants) | 38
Number analyzed (Chemotherapy Expected) | 152
Number of Chemotherapy cycles | 123

5. Secondary Outcome: Neurotoxicity
Description: Total number of patients with neurotoxic events during treatment
Time Frame: 2-year
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose Sequential Chemoimmunotherapy
Number analyzed (Participants) | 38
Participants | 2

ADVERSE EVENTS:
Time Frame: 5 years
Description: Serius
Groups:
- High-dose Sequential Chemoimmunotherapy: Two courses of methotrexate 3.5 g/mq day 1 and cytarabine 2 g/mq twice a day, for two days, Rituximab 375 mg/mq days 3 & 11 and Intrathecal liposomal cytarabine 50 mg day 6(Ph I) followed in case of response by cyclophosphamide 7 g/mq plus Rituximab 375 mg/mq and Intrathecal liposomal cytarabine 50 mg Leukapheresis A and cryopreservation (Ph II), Cytarabine 2 g/mq twice a day for 4 days, Rituximab 375 mg/m2 and Reinfusion of stem cells (Phase III), etoposide 2 g/mq, Intrathecal liposomal cytarabine 50 mg (Ph IV) and high-dose Thiotepa-BCNU supported by autologous stem cell transplant (Phase V), and whole-brain radiotherapy in patients who do not achieve a complete remission after chemotherapy (Phase VI)
  High-dose sequential chemotherapy and autologous transplant: Two courses of methotrexate 3.5 g/mq day 1 and cytarabine 2 g/mq twice a day, for two days, Rituximab 375 mg/mq days 3 & 11 and Intrathecal liposomal cytarabine 50 mg day 6(Phase I) followed in case of response by cyclophosphamide 7 g/mq plus Rituximab 375 mg/mq and Intrathecal liposomal cytarabine 50 mg Leukapheresis A and cryopreservation (Phase II), Cytarabine 2 g/mq twice a day for 4 days, Rituximab 375 mg/m2 and Reinfusion of stem cells (Phase III), etoposide 2 g/mq, Intrathecal liposomal cytarabine 50 mg (Phase IV) and high-dose Thiotepa-BCNU supported by autologous stem cell transplant (Phase V), and whole-brain radiotherapy in patients who do not achieve a complete remission after chemotherapy (Phase VI)
Arm/Group | High-dose Sequential Chemoimmunotherapy
All-Cause Mortality (participants affected / at risk) | 22/38
Serious Adverse Events (participants affected / at risk) | 4/38
Other Adverse Events (participants affected / at risk) | 3/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-dose Sequential Chemoimmunotherapy (N=38)
death (Blood and lymphatic system disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-dose Sequential Chemoimmunotherapy (N=38)
febril neutropenia (General disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes